CLINICAL TRIAL: NCT07057063
Title: Effect of Light Therapy on Pain and Synovitis in Patients With Knee Synovitis: Study Protocol for a Randomized Controlled Trial
Brief Title: Light Therapy on Pain and Synovitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, FU Siu Ngor, Peter Hung Professor in Pain Management, Assoc. Head(RS), ADoRISports & Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20230214003 PolyU
Record Dates: First submitted 2025-06-25; First posted 2025-07-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Knee Pain Chronic; Synovitis of Knee; Light Therapy
Keywords: Light therapy; Photobiomodulation; Chronic knee pain; Synovitis; Randomized controlled trial; Non-pharmacological intervention; physical therapy
MeSH Terms: conditions — Synovitis | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation will be not revealed to the participants and ultrasound assessors until the completion of the final data analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 810 nm Light Therapy Group (Experimental): Participants receive 810 nm light therapy using a wearable device, twice per week for 5 weeks.
  Interventions: Device: 810 nm Light Therapy
- Sham Therapy Group (Placebo Comparator): Participants receive sham therapy with the same device that emits no therapeutic light, twice per week for 5 weeks.
  Interventions: Device: Sham Light Therapy

INTERVENTIONS:
Device: 810 nm Light Therapy — Light therapy at 810 nm, 39 J/cm², delivered via wearable device.
  Arms: 810 nm Light Therapy Group
Device: Sham Light Therapy — Identical device, no light output, delivered via wearable device.
  Arms: Sham Therapy Group

SUMMARY:
Background: Knee pain is a common complaint among middle-aged and older adults, often leading to reduced mobility and diminished quality of life. Synovitis is a major underlying cause, present in up to 80% of individuals with moderate knee pain. While light therapy has shown anti-inflammatory and analgesic effects in preclinical studies, our prior animal experiments revealed that light therapy at 810 nm significantly alleviated inflammation and pain-like behaviors. These findings suggest a potential wavelength-specific therapeutic effects. However, it remains unclear whether such effects can be replicated in humans. This study aims to evaluate the efficacy of 810 nm light therapy, compared to sham treatment, in reducing knee pain and synovitis in patients with chronic knee pain and knee synovitis.

Methods/design:

This is a randomized, placebo-controlled clinical trial involving 90 participants with chronic knee pain and ultrasound-detected synovitis. Participants will be randomized into two groups to receive 810 nm light therapy, or sham therapy, delivered twice weekly over five weeks. Primary outcomes include knee pain assessed by the Visual Analogue Scale (VAS) and synovitis assessed by ultrasound. Secondary outcomes include the Knee injury and Osteoarthritis Outcome Score (KOOS), the 30-second chair stand test, and the 40-meter fast-paced walk test. Outcome assessments will be performed at baseline, post-intervention (week 5), and at 1 month and 6 months after treatment completion. Linear mixed-effects models will be used to compare outcome changes between groups.

Discussion:

This trial will assess whether 810 nm light therapy provides clinically meaningful benefits for reducing knee pain and synovitis in humans, building on promising preclinical findings. Results from this study may support the use of near-infrared light as a safe, non-invasive, and effective intervention for synovitis-related knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 40 and 80 years
* Able to provide written informed consent
* Have experienced knee pain that persists or recurs for more than 3 months
* A knee pain score of at least 30 mm on the 100-mm Visual Analogue Scale (VAS) during the past week
* Ultrasound-measured knee synovitis ≥1
* Presence of knee OA according to criteria established by the American College of Rheumatology

Exclusion Criteria:

* Anticipated need for knee surgery within the next one year
* Previous or planned knee replacement within the next one year
* Knee surgery or other physical therapy in the previous 3 months
* Use of intra-articular, intra-muscular, or oral corticosteroids in previous 4 weeks
* Malignant tumors or other life-threatening diseases
* Severe mental disorders, including but not limited to schizophrenia, bipolar disorder, or major depressive disorder, that may interfere with the participant's ability to comply with the study protocol or provide informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Knee pain (Visual Analogue Scale, VAS) | Baseline, Week 5, 1-month follow-up, 6-month follow-up
  Knee pain severity will be assessed using a 100-mm Visual Analogue Scale (VAS), based on average pain over the past week.
Knee synovitis grade (Ultrasound assessment) | Baseline, Week 5, 1-month follow-up, 6-month follow-up
  Knee ultrasound will be performed by an ultrasound physician with over 8 years of experience, following the published protocol (Bruyn GAW, Naredo E, Damjanov N, et al (2016) An OMERACT reliability exercise of inflammatory and structural abnormalities in patients with knee osteoarthritis using ultrasound assessment. Ann Rheum Dis 75:842-846. https://doi.org/10.1136/ann). The items measured included the maximal score for synovitis obtained at the suprapatellar or parapatellar recesses, with a range of 0-3. Grade 0 indicates no synovitis; Grade 1 represents minimal distension of the recess by abnormal internal hypoechoic or anechoic material (relative to subdermal fat tissue); Grade 2 signifies moderate distension or enlargement of the recess by abnormal internal hypoechoic or anechoic material with a flat or concave superficial limit; and Grade 3 denotes severe distension or enlargement of the recess by abnormal internal hypoechoic or anechoic material with a bulging superficial limit.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Score (KOOS) | Baseline, Week 5, 1-month follow-up, 6-month follow-up
  Knee Injury and Osteoarthritis Score (KOOS) that includes subdomains of pain (9 items), other symptoms (7 items), function and daily living (short PS version 7 items), and knee-related quality of life (4 items) will be used in this study. A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Lower limb function (30-second chair stand test) | Baseline, Week 5, 1-month follow-up, 6-month follow-up
  A standard chair without arms will be used for the chair stand test (Dobson F, Bennell KL, Hinman RS, et al (2013) Recommended performance based tests to assess physical function in patients with hip/knee OA. Osteoarthr Cartil 8:1042-52). Participants will begin the test seated with their arms crossed over their chest. They will be instructed to stand up fully, so hips and knees are fully extended, and return to the seated position as many times as possible within 30 seconds, while keeping their arms crossed. The total number of chair stands (up and down equals one stand) completed in 30 seconds will be recorded. If a full stand has been completed at 30 seconds (i.e. standing fully erect or on the way down to the sitting position), then this final stand is counted in the total.
Walking speed (40-meter fast-paced walk test) | Baseline, Week 5, 1-month follow-up, 6-month follow-up
  The 40-meter walk test will be conducted on a marked 10-meter walkway, with cones placed 2 meters beyond each end to facilitate turning. Participants wore comfortable walking footwear. After a brief practice trial to ensure understanding, participants will be instructed to walk as quickly and safely as possible, without running, along the walkway. They turned around the cones at each end and repeated the process until completing a total distance of 40 meters, involving three turns. Timing started when participants began walking and stopped when they crossed the start line after completing the full distance. Walking speed (m/s) will be calculated by dividing 40 meters by the recorded time (Dobson F, Bennell KL, Hinman RS, et al (2013) Recommended performance based tests to assess physical function in patients with hip/knee OA. Osteoarthr Cartil 8:1042-52).
Adverse events monitoring for light therapy | Throughout the intervention period and at all follow-up visits (up to 6 months)
  Participants will be closely monitored for adverse events (AEs) at each treatment and visit throughout the study. If any AEs occur (e.g., cutaneous irritation, redness, or itching at the treatment site), they will be documented on a separate form and reported to the principal investigators (PIs) within 24 hours. This monitoring will ensure that any adverse events are promptly addressed and that the safety of participants is prioritized throughout the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Buji Community Service Center, Longgang District, Shenzhen, China
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article, after de-identification, will be shared. Data will be available upon reasonable request from qualified researchers, subject to ethics approval and data use agreement. The data will become available after the publication of the main results and will be accessible for a period of 5 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and supporting documents will be available beginning 6 months after publication of the primary results, and will be available for 5 years thereafter.
Access Criteria: Data will be available to qualified researchers whose proposed use of the data has been approved by an independent review committee. Access will be provided after signing a data access agreement. Interested researchers should contact the Principal Investigator by email.

REFERENCES:
- [Background] 1. Duong V, Oo WM, Ding C, et al (2023) Evaluation and Treatment of Knee Pain: A Review. Jama 330:1568-1580. https://doi.org/10.1001/jama.2023.19675 2. Baker K, Grainger A, Niu J, et al (2010) Relation of synovitis to knee pain using contrast-enhanced MRIs. Ann Rheum Dis 69:1779-83. https://doi.org/10.1136/ard.2009.121426 3. Blom AB, van Lent PLEM, Holthuysen AEM, et al (2004) Synovial lining macrophages mediate osteophyte formation during experimental osteoarthritis. Osteoarthr Cartil 12:627-35. https://doi.org/10.1016/j.joca.2004.03.003 4. Mathiessen A, Conaghan PG (2017) Synovitis in osteoarthritis: Current understanding with therapeutic implications. Arthritis Res Ther 19:1-9. https://doi.org/10.1186/s13075-017-1229-9 5. Zhu Z, Li J, Ruan G, et al (2018) Investigational drugs for the treatment of osteoarthritis, an update on recent developments. Expert Opin Investig Drugs 27:881-900. https://doi.org/10.1080/13543784.2018.1539075 6. Mussttaf RA, Jenkins DFL, Jha AN (2019) Assessing the impact of low level laser therapy (LLLT) on biological systems: a review. Int J Radiat Biol 95:120-143. https://doi.org/10.1080/09553002.2019.1524944 7. de Freitas LF, Hamblin MR (2016) Proposed Mechanisms of Photobiomodulation or Low-Level Light Therapy. IEEE J Sel Top Quantum Electron 22:. https://doi.org/10.1109/JSTQE.2016.2561201 8. de Oliveira VLC, Silva JA, Serra AJ, et al (2017) Photobiomodulation therapy in the modulation of inflammatory mediators and bradykinin receptors in an experimental model of acute osteoarthritis. Lasers Med Sci 32:87-94. https://doi.org/10.1007/s10103-016-2089-2 9. Hagiwara S, Iwasaka H, Okuda K, Noguchi T (2007) GaAlAs (830 nm) low-level laser enhances peripheral endogenous opioid analgesia in rats. Lasers Surg Med 39:797-802. https://doi.org/10.1002/lsm.20583 10. dos Santos SA, dos Santos Vieira MA, Simões MCB, et al (2017) Photobiomodulation therapy associated with treadmill training in the oxidative stress in a collagen-induced arthrit